CLINICAL TRIAL: NCT01347931
Title: In-home Evaluation of the Breathe Technologies Noninvasive Open Ventilation (NIOV™) System in Patients With Severe Respiratory Insufficiency
Brief Title: In-home Evaluation of a Noninvasive Open Ventilation System in Patients With Severe Respiratory Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Breathe Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP-00-0034
Record Dates: First submitted 2011-05-03; First posted 2011-05-05 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Airflow Obstruction, Chronic; Chronic Obstructive Airway Disease; Chronic Obstructive Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Oxygen Inhalation Therapy; Cannula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIOV System (Experimental): Noninvasive ventilation and oxygen delivered via NIOV System oxygen using an open nasal interface. Connected to standard portable oxygen cylinder
  Interventions: Device: NIOV System
- Standard Oxygen Therapy (Active Comparator): Supplemental oxygen using standard oxygen cannula connected to a portable oxygen cylinder.
  Interventions: Device: Standard Oxygen Cannula

INTERVENTIONS:
Device: NIOV System — Each subject's standard oxygen therapy will be used as the control treatment and compared to the test ventilator (NIOV) system during selected activities of daily living.
  Other Names: NIOV; Oxygen; O2
  Arms: NIOV System
Device: Standard Oxygen Cannula — Supplemental oxygen via a standard oxygen cannula connected to a portable oxygen cylinder
  Other Names: Cannula
  Arms: Standard Oxygen Therapy

SUMMARY:
The Breathe NIOV™ System will reduce the work of breathing in subjects with chronic respiratory insufficiency who require long-term oxygen therapy (LTOT). The Breathe system will accomplish this by providing oxygen under pressure and augmenting the subject's spontaneous tidal volumes. The combination of efficient oxygen delivery, assisted ventilation, and a comfortable low-profile device, will result in a mean improvement in perceived well-being and ability to perform ADLs, as measured by patient-reported outcome (PRO) instruments.

DETAILED DESCRIPTION:
This will be a prospective, open-label, crossover study in up to 12 stable subjects with chronic respiratory insufficiency who require LTOT. Each subject's standard oxygen therapy will be used as the control treatment and compared to the test ventilator system during selected activities of daily living. Subjects will participate in the study for up to 9 home visits, with Visits 1 and 2 each lasting for approximately 4 hours, and Visits 3-9 lasting approximately 1-2 hours each. Subjects may discontinue study participation at any time.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects, 21-80 years of age
* Diagnosis of chronic respiratory insufficiency including COPD and interstitial lung disease
* Requires use of continuous nasal oxygen of at least 2 lpm
* Reports limitation of activity due to fatigue or breathlessness
* Fluent in written and spoken English language
* Ability to be properly fitted with the Breathe nasal mask
* Ability to tolerate and be appropriately titrated on the Breathe ventilator
* Ability to communicate self-assessment of dyspnea, comfort, and fatigue
* Ability and willingness to participate in the study including walking and other activities of daily living
* Ability to provide written informed consent

Exclusion Criteria:

* Recent history of frequent or severe epistaxis
* Symptoms of acute respiratory exacerbation within 48 hours of Study Day 1
* Discharge from the hospital within 30 days of study enrollment
* Subjects, who in the opinion of the Investigator, are not suitable candidates for enrollment or who are unlikely to be able to comply with trial requirements
* Subjects with conditions that, in the Investigator's opinion, contraindicates study participation

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian W Carlin, MD, Principal Investigator — West Penn Allegheny Health System
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Oxygen Therapy: Supplemental oxygen delivered via standard nasal cannula connected to a portable oxygen cylinder.
  Breathe NIOV System: Each subject's standard oxygen therapy will be used as the control treatment and compared to the test ventilator (NIOV) system during selected activities of daily living.
Period: Standard Oxygen Therapy
Arm/Group | Standard Oxygen Therapy
Started | 30
Completed | 29
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: NIOV System
Arm/Group | Standard Oxygen Therapy
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Per protocol
Groups:
- Overall Study Group: All subjects participating in 2-way crossover design study
Arm/Group | Overall Study Group
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Activity Endurance Time
Description: Time in minutes of sustained activity while using test treatments
Time Frame: Measured during single day study visit
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Standard Oxygen Therapy: Supplemental oxygen delivered via standard nasal cannula connected to a portable oxygen cylinder.
  NIOV System: Each subject's standard oxygen therapy will be used as the control treatment and compared to the test ventilator (NIOV) system during selected activities of daily living.
- Breathe NIOV System: Noninvasive ventilation delivered via NIOV System oxygen using an open nasal interface. Connected to standard portable oxygen cylinder
  NIOV System: Each subject's standard oxygen therapy will be used as the control treatment and compared to the test ventilator (NIOV) system during selected activities of daily living.
Arm/Group | Standard Oxygen Therapy | Breathe NIOV System
Number analyzed (Participants) | 29 | 29
minutes | 7.24 (5.21) | 13.38 (7.50)
Statistical Analysis 1: Comparison: Standard Oxygen Therapy vs Breathe NIOV System; A sample size of 26 patient pairs was determined based on the assumption of a true treatment difference in mean ADL endurance time of 4 ± 7 minutes using a two-tailed, paired t test (α=0.05, power=0.80); Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 4, 95% CI 2-sided [2 to 10], Standard Deviation 7

2. Secondary Outcome: Arterial Oxygen Saturation
Description: O2 saturation measured by pulse oximetry
Time Frame: Measured during activity testing in a single day study visit
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: percentage of oxyHb saturation
Arm/Group | Standard Oxygen Therapy | Breathe NIOV System
Number analyzed (Participants) | 29 | 29
percentage of oxyHb saturation | 90.65 (4.87) | 94.78 (1.99)
Statistical Analysis 1: Comparison: Standard Oxygen Therapy vs Breathe NIOV System; Two-tailed t test; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 3, 95% CI 2-sided [1 to 7], Standard Deviation 4

3. Secondary Outcome: Borg Dyspnea Score
Description: Borg Dyspnea score is measured using a 11-point visual analog scale. The lower the score on the scale, the less breathlessness patient experiences. The score ranges from:
  0 = No breathlessness at all, representing better outcome 10 = Maximum, representing worse outcome
Time Frame: Measured during activity testing in a single day study visit
Population: Per Protocol
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Standard Oxygen Therapy | Breathe NIOV System
Number analyzed (Participants) | 29 | 29
units on a scale | 3 [2.80 to 4.07] | 1 [1.00 to 2.40]

ADVERSE EVENTS:
Time Frame: Continuously monitored during a Single day study visit lasting up to 4 hours
Arm/Group | Standard Oxygen Therapy | Breathe NIOV System
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No